CLINICAL TRIAL: NCT00523159
Title: Phase 2, Randomized, Open Label, Multicenter Study of Intradermal IMA901 Plus GM-CSF With or Without Low Dose Cyclophosphamide Pre-treatment in Advanced Renal Cell Carcinoma Patients With Measurable Disease
Brief Title: IMA901 in Advanced Renal Cell Carcinoma Patients With Measurable Disease
Acronym: IMA901-202
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immatics Biotechnologies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT Nr: 2006-006370-25
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2010-02

CONDITIONS: Renal Cell Carcinoma
Keywords: clear cell renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Pre-treatment with a single low dose of Cyclophosphamide followed by IMA901 vaccination plus GM-CSF as adjuvant
  Interventions: Drug: Endoxana, IMA901, Leukine
- 2 (Other): No pre-treatment with Cyclophosphamide before vaccination with IMA901 and GM-CSF as adjuvant
  Interventions: Drug: IMA901 and Leukine

INTERVENTIONS:
Drug: Endoxana, IMA901, Leukine — a single i.v. infusion of Cyclophosphamid and then patients received vaccination therapy with intradermal (i.d.) injections of GM-CSF followed by i.d. injections of IMA901
  Arms: 1
Drug: IMA901 and Leukine — Intradermal injection of GM-CSF followed by intradermal injection of IMA901
  Arms: 2

SUMMARY:
This study was conducted in order to evaluate the efficacy and safety of the cancer vaccine IMA901 and GM-CSF as adjuvant in the treatment of advanced renal cell carcinoma.

Patients received vaccination with GM-CSF followed by IMA901 during the study period of 9 months. Patients received pre-treatment with a single i.v. infusion of cyclophosphamide prior to the first vaccination.

DETAILED DESCRIPTION:
This is a multicenter, open label, randomized phase 2 study which investigated the effect of a second-line systemic treatment with IMA901 plus GM-CSF in RCC patients. Randomization was done according to a pre-treatment with low-dose cyclophosphamide (CY). Secondary endpoints comprised tumor response parameters.

The study population consisted of HLA-A*02-positive men or women with advanced RCC of the clear-cell type classified as having a favorable or intermediate risk after first-line systemic therapy for. Patients had to be aged 18 years or older, had at least have one measurable tumor lesion and had have received first-line tyrosine kinase inhibitor or cytokine systemic therapy for advanced disease, during or after which the patient had experienced disease progression.

Patients in both arms received a total of 17 vaccinations with GM-CSF followed by IMA901 during the 9 month treatment period.

At screening baseline tumor status was assessed by CT or MRI. During the study tumor assessments were performed every 6 weeks.

Immunomonitoring (T-cell responses to peptides contained in IMA901 and analysis of other immune cell populations that may influence T-cell responses), serum levels of antibodies and molecules with suspected influence on immune response were assessed on several occasions during the study.

Safety assessment comprised continuous adverse event reporting, regular physical examinations and regular assessments of vital signs, hematology, blood chemistry and urine. A 12-lead ECG was performed at screening and at the end of the study. Pregnancy testing was performed according to applicable legislation in the country where the trial was performed. At the very least, women of childbearing potential had have to undergo a pregnancy test during screening for the study, before the first dose was applied and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years
* HLA type: HLA-A*02-positive
* Histologically documented advanced clear-cell RCC
* Patients who have received first-line tyrosine kinase inhibitor or cytokine systemic therapy for advanced disease systematic therapy for advanced disease and must be candidates for second-line therapy (NOTE: in Germany and Austria only patients after first-line tyrosine kinase inhibitor failure will be included into the study)
* Patients having experienced documented tumor progression
* At least one unidimensional measurable target lesion
* Karnofsky Performance Status ≥ 80%
* Favorable or intermediate risk according to the 3-score MSKCC criteria.
* Able to understand the nature of the study and give written informed consent
* Willingness and ability to comply with the study protocol for the duration of the study

Exclusion Criteria:

* Poor risk according to the 3-score MSKCC criteria
* Immunosuppressive therapy within 4 weeks before study entry, e.g. corticosteroid treatment
* History of other malignant tumors, except non-melanoma-skin cancer or curatively excised cervical carcinoma in situ
* Presence of brain metastases on MRI or CT scan
* Patients with a history or evidence of systemic autoimmune disease
* Any vaccination in the two weeks before study entry
* Any planned prophylactic vaccination from study entry until the end of the induction period (5 weeks after the first vaccination)
* Known active hepatitis B or C infection
* Known HIV infection
* Any other infection with a biological agent that can cause a severe disease and poses a severe danger to lab personnel working on patient tissues.
* Any of the following in the 4 weeks before study entry:

  1. Major surgery
  2. Anticancer treatments including (but not limited to) cytotoxic chemotherapy, radiotherapy, immunotherapy, hormone therapy, tyrosine kinase inhibitors, monoclonal antibodies
  3. Unresolved toxicity from prior anticancer treatments including (but not limited to) cytotoxic chemotherapy, hormone therapy, tyrosine kinase inhibitors, monoclonal antibodies, radiotherapy, or immunotherapy
  4. Received study drug within any clinical study
* Any of the following abnormal laboratory values:

  1. Hematology: Hb < 9 g/dL; WBC < 3 x 109/L; neutrophils < 1.5 x 109/L; lymphocytes < 1.0 x 109/L; platelets < 100 x 109/L
  2. Liver function: serum bilirubin > 1.5 x upper normal limit (unless a history of Gilbert's disease); ALAT or ASAT > 3 x upper normal limit (>5 x upper normal limit if liver metastases are present)
  3. Renal function: serum creatinine > 200 µmol/L
* Patients with other significant diseases currently uncontrolled by treatment which might interfere with study completion, for example:

  1. Heart failure or non compensated active heart disease
  2. Severe coronary heart disease, cardiac arrhythmia requiring medication, or uncontrolled hypertension
  3. Symptomatic neurotoxicity (motor or sensory) ≥ grade 2 National Cancer Institute - Common Toxicity Criteria (NCI-CTC).
  4. Severe pulmonary dysfunction
* Psychiatric disabilities, seizures or central nervous system disorders that may interfere with the ability to give informed consent or perform adequate follow-up in the investigator's opinion
* Active infections requiring oral or intravenous antibiotics
* Women or men who decline to practice a medically approved method of contraception
* Pregnancy or breastfeeding
* Any condition which in the judgment of the investigator would place the patient at undue risk or interfere with the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Disease control rate | after 26 weeks

SECONDARY OUTCOMES:
Tumor response rates and SD rate | after 26 and 38 weeks
Duration of response | from the time response is first documented until the first date of recurrence or PD
Time to response | From Visit c to PR or CR
TTP | From visit C to until tumor progression
PFS and OS | From visit C to tumor progression or death
DCR | after 38 weeks on study
Immune response | Visit C, 1, 5, 6, 7, 10 and 14
Effect of cyclophosphamide pre-treatment on immune response | Visit C, 1, 5,6,7, 10, 14
Safety | From inclusion on the study until 3 weeks after end of study visit

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kirner, PhD, Study Director — Immatics Biotechnologies GmbH
Locations (44):
- Medizinische Universität Salzburg - Universitätsklinik für Innere Medizin III, Salzburg, Austria
- Bulgaria (2):
  - National Oncology Hospital - Urology, Sofia
  - Regional Oncodispensary with inpatient sector-Sofia District, Sofia
- Germany (13):
  - Charité Campus Mitte-Klinik für Urologie, Berlin
  - Charité Campus Benjamin Franklin - Medizinische Klinik III, Berlin
  - Zeisigwaldkliniken Bethanien Chemnitz GmbH, Chemnitz
  - Universitätsklinikum Essen, Essen
  - Klinik der Johann-Wolfgang-Goethe-Universität, Frankfurt am Main
  - Universitätsklinikum Hamburg-Eppendorf Onkologisches Zentrum (Onkologie / Hämatologie), Hamburg
  - Universitätsklinikum Heidelberg - Klinik für Urologie, Heidelberg
  - Universitätsklinikum Schleswig Holstein - Campus Lübeck, Lübeck
  - Universitätsklinikum Mainz - 3. Medizinische Klinik, Mainz
  - Klinikum der Universität - München Großhadern, Munich
  - Urologische Klinik Dr. Castringius - München-Planegg, Planegg
  - Universitätsklinikum Tübingen - Klinik für Urologie, Tübingen
  - Schwarzwald-Baar-Klinik - Abt. Hämatologie und Onkologie, Villingen-Schwenningen
- Hungary (9):
  - DRC Gyógyszervizsgáló Központ Kft, Balatonfüred
  - Semmelweis Egyetem - Urológiai Klinika, Budapest
  - Bajcsy-Zsilinszky Kórház - Urológia Osztály, Budapest
  - Fövárosi Önk.Szt.Imre Kórház - Belgyógyászat-Kliniko-FFarmakológia, Budapest
  - Országos Onkológiai Intézet - Kemoterápia C osztály-Klinikofarmakológia, Budapest
  - Debreceni Egyetem Orvos és Egészségtudományi Centrum, Debrecen
  - Hajdú-Bihar Megyei Önk. Kenézy Gyula Kórház/Urológia Osztály, Debrecen
  - BAZ megyei Kórház - Urológia Osztály, Miskolc
  - Pécs Orvostudomanyi Egyetem - Urológiai Klinika, Pécs
- Poland (3):
  - Klinika Chemioterapii Nowotworow - Uniwersytetu Medycznego, Lodz
  - Klinika Onkologii Wojskowego Institutu Medycznego, Warsaw
  - Clinic of Urology and Urological Oncology Medica University Hospital, Wroclaw
- Romania (4):
  - Oncology Institute "Prof. Dr. Alexandru Trestioreanu", Bucharest
  - Oncology Institute - "Prof. Dr. Alexandru Trestioreanu", Bucharest
  - Oncology Institute "Prof. Dr. Ion Chiricuta", Cluj-Napoca
  - Clinical County Hospital Oradea, Oradea
- Slovakia (4):
  - National Cancer Institut - "Narodny onkologicky ustav", Bratislava
  - Clinic of Radiotherapy and Oncology - East Slovak Oncology Institute, Košice
  - Martin Faculty Hospital, Martin
  - Department of Clinical Oncology - Faculty Hospital with Policlinic of J.A. Reiman, Prešov
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital 12 de Octubre, Madrid
  - Clinica Universitaria de Navarra - Servicio de Oncologia, Pamplona
- University Hospital - Medicine Oncology, Geneva, Switzerland
- United Kingdom (3):
  - Beatson Oncology Centre, Glasgow
  - Christie Hospital NHS Trust, CRUK Department of Medical Onkology - Paterson Institute for Cancer Research, Manchester
  - University of Surrey - Postgraduate Medical School, Surrey